CLINICAL TRIAL: NCT03198728
Title: A 12-Month, Randomized, Active-controlled, Open-label Study of the Efficacy and Safety of Oral Testosterone Undecanoate in Hypogonadal Men (RE-TUne)
Brief Title: Efficacy and Safety of Oral Testosterone Undecanoate in Hypogonadal Men
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Marius Pharmaceuticals (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MRS-TU-2019
Record Dates: First submitted 2017-06-21; First posted 2017-06-26 (Actual); Results first posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Hypogonadism, Male
MeSH Terms: conditions — Eunuchism | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant
Masking Description: Open label
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SOV2012-F1-treated (Experimental): 200 patients treated with SOV2012-F1, starting dose of 600 mg - (400 mg with morning meal and 200 mg with evening meal). Dose titrated on Days 28 and 56 up to a maximum of 600 mg TU in the morning and 400 mg in the evening or down to 200 mg TU in the morning based on plasma T at Days 14 and 42.
  Interventions: Drug: SOV2012-F1
- Andro-Gel™ treated (Active Comparator): 100 patients treated with AndroGel, starting dose of 40.5 mg QD. Dose titrated according to approved label, using samples from Days 14 and 42 and dose adjustments on Days 28 and 56.
  Interventions: Drug: AndroGel

INTERVENTIONS:
Drug: SOV2012-F1 — oral preparation of testosterone undecanoate (TU)
  Arms: SOV2012-F1-treated
Drug: AndroGel — topical testosterone gel 1.62%
  Arms: Andro-Gel™ treated

SUMMARY:
This will be a randomized, multicenter, open-label, active-controlled, efficacy, and safety study in adult hypogonadal men. The study duration is 12 months (365 days), including a 90-day, open-label efficacy period and a 9-month (275-day) safety evaluation period.

DETAILED DESCRIPTION:
MRS-TU-2019 was a 12-month study designed to determine the efficacy of oral SOV2012-F1 as measured by the percentage of male hypogonadal subjects with average total testosterone (T Cavg) in plasma within the normal range after 90 days of treatment. This study included an AndroGel™ arm as a safety comparator; after the 90-day efficacy period, dosing continued for 9 additional months in both arms to gather safety data. This study also examined the percentage of SOV2012-F1-treated subjects with maximum total testosterone (Cmax) in plasma values after 90 days of treatment: a. ≤1.5 X upper limit of normal (ULN); b. 1.8 X ULN to 2.5 X ULN' and c. >2.5 X ULN. The study also included an adrenal cortical function substudy conducted in 30 SOV2012-F1 subjects and 15 AndroGel subjects. Four patient-reported outcome measures were also used during the study: IPSS, PDQ, SF-36 and IIEF.

ELIGIBILITY:
Inclusion Criteria:

1. Male aged 18 to 65 years, inclusive, at the time of providing informed consent to participate in the study.
2. Hypogonadism defined as having 2 consecutive serum total T levels≤ 281 ng/dL based on a blood sample, drawn at least 3 days apart, between 7 a.m. and 10 a.m.
3. At least 1 clinical feature consistent with male hypogonadism. If a subject is receiving commercial TRT prior to Screening Visit 1, he must have a history of at least 1 clinical feature consistent with male hypogonadism.
4. Must be naïve to androgen replacement therapy or washed out adequately of prior androgen replacement therapies; willing to cease current T treatment; or currently not taking any T treatment. Subjects must remain off all forms of T, except for dispensed study drug, throughout the entire study.
5. No unstable ongoing concomitant medical conditions. Treated and well-controlled conditions such as type 2 diabetes, hypertension, or dyslipidemia are acceptable with stable medication in place for at least 3 months prior to study entry:

   1. Hemoglobin A1c ≤ 8.0%
   2. BP < 150/90 mm Hg
   3. Low-density lipoprotein cholesterol < 190 mg/dL.
6. Subjects with an endocrine disorder requiring treatment other than hypogonadism must be on a stable dose of replacement medication for at least 3 months prior to study entry.
7. Adequate venous access to allow collection of a number of blood samples via a venous cannula.
8. Written informed consent to participate in the study and ability to comply with all study requirements.

Exclusion Criteria:

1. Serum PSA > 2.5 ng/ml and/or abnormal prostate gland on palpation, eg, palpable nodes, at Screening Visit 2.
2. Received oral, topical, intranasal, or buccal T therapy within the previous 2 weeks, intramuscular T injection of short-acting duration within the previous 4 weeks, intramuscular T injection of long-acting duration within the previous 20 weeks, or T implantable pellets within the previous 6 months.
3. Use of any drug that could interfere with measurement or assessment of serum androgen levels, including 5 alpha-reductase inhibitors, anabolic steroids, and drugs with antiandrogenic properties (eg, spironolactone, cimetidine, flutamide, bicalutamide, and ketoconazole). These drugs must be stopped for at least 1 month prior to study entry (6 months in the case of dutasteride). Patients taking potent, long-acting opiate therapy on a daily basis are not eligible for the study. Conversely, ad hoc use of potent, short-acting opiates for a period of less than 7 days may be permitted after discussion with the Marius Pharmaceuticals medical monitor.
4. Use of over-the-counter products, including natural health products (eg, food supplements and herbal supplements such as saw palmetto or phytoestrogens) that may affect total T levels, within 7 days prior to study entry.
5. History of drug or alcohol abuse within the past 2 years that in the opinion of the investigator could interfere with study participation and/or influence study efficacy and safety endpoints assessments.
6. Unstable or chronic disease that could interfere with participation in the study or patient safety, including psychiatric disorders.
7. Myocardial infarction, coronary artery surgery, heart failure, stroke, unstable angina, or other unstable cardiovascular disease within the past 6 months.
8. Abnormal ECG considered clinically significant by investigator at Screening.
9. Diagnosis of any cancer within the previous 5 years other than basal or squamous cell skin cancer with clear margins.
10. Any surgical or medical condition that might alter administration of the study drug or comparator, including history of gastric surgery, cholecystectomy, vagotomy, bowel resection, or any surgical procedure that might interfere with gastrointestinal motility, pH, or absorption of TU.
11. Duodenal or gastric ulcers, or gastrointestinal/rectal bleeding during the 3 months prior to screening.
12. Chronic skin conditions on the chest or upper arms that would prevent administration of AndroGel in a manner designed to ensure reliable and consistent absorption thereof.
13. Human immunodeficiency virus (HIV) infection.
14. Chronic hepatitis B virus and/or hepatitis C virus (HCV) infection (as determined by positive testing for hepatitis B virus surface antigen or HCV antibody with confirmatory testing, ie, detectable serum HCV ribonucleic acid [RNA]).
15. Clinically significant abnormal laboratory values at screening including but not limited to:

    1. Elevated liver enzymes (aspartate aminotransferase [AST], alanine aminotransferase [ALT] > 2x upper limit of normal)
    2. Estimated glomerular filtration rate < 60 ml/min/1.73m2 as calculated by the Modification of Diet in Renal Disease formula
    3. Hemoglobin < 11.0 g/dL or > 16.0 g/dL. For a subject previously on testosterone replacement therapy with less than 30 days washout prior to screening Visit 2, hemoglobin < 11.0 g/dL or > 17.0 g/dL.
16. Severe and untreated obstructive sleep apnea syndrome.
17. Severe lower urinary tract symptoms (American Urological Association/ IPSS ≥ 19).
18. History of any clinically significant illness, infection, or surgical procedure within 1 month prior to study entry.
19. Past, current, or suspected prostate or breast cancer.
20. History of long QT syndrome or unexplained sudden death in a first-degree relative (parent, sibling, or child).
21. Concurrent treatment with medications that may impact the absorption, distribution, metabolism, or excretion of TU or place the subject at risk for treatment with T.
22. Subject has a partner who is currently pregnant or planning pregnancy during the course of the study.
23. Treatment with any other investigational drug within 30 days of study entry or > 5 half-lives (whichever is longer) and at any time during the study.
24. History of noncompliance to medical regimens or potential unreliability in the opinion of the investigator.
25. Unwilling or unable to comply to the dietary requirements for this study.
26. History of polycythemia, either idiopathic or associated with TRT.
27. Donated blood (≥ 500 mL) within the 12-week period prior to study entry.
28. History of an abnormal bleeding tendency or thrombophlebitis within the previous 2 years that is not linked to venipuncture or intravenous cannulation.
29. Onset of gynecomastia within the previous 6 months.
30. For adrenocorticotropic hormone (ACTH) stimulation substudy only: Primary or secondary adrenal insufficiency.
31. For Bioanalytical Sample Stability Substudy only: subjects with a hemoglobin less than 13 g/dL at most recent assessment* [should be excluded].

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 314 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alastair Smith, MB, ChB, Study Director — Syneos Health; Om Dhingra, PhD, Study Chair — Marius Pharmaceuticals
Locations (36):
- United States (36):
  - Central Research Associates, Inc., Birmingham, Alabama
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Quality of Life Medical and Research Centers, LLC, Tucson, Arizona
  - San Diego Sexual Medicine, San Diego, California
  - South Florida Medical Research, Aventura, Florida
  - PAB Clinical Research, Brandon, Florida
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Jacksonville Impotence Treatment Center, Jacksonville, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Meridien Research, Lakeland, Florida
  - My Community Research Center, Miami, Florida
  - Oviedo Medical Research, LLC, Oviedo, Florida
  - Meridien Research, St. Petersburg, Florida
  - Primary Care Research Group, Atlanta, Georgia
  - Northwest Clinical Trials, Boise, Idaho
  - Advanced Clinical Research, Meridian, Idaho
  - Central Kentucky Research Associates, Lexington, Kentucky
  - Centex Studies, Inc., Lake Charles, Louisiana
  - Men's Health Boston, Chestnut Hill, Massachusetts
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - Palm Research Center, Inc., Las Vegas, Nevada
  - Accumed Research Associates, Garden City, New York
  - Manhattan Medical Research Practice, PLLC, New York, New York
  - Rapha Institute For Clinical Research, Fayetteville, North Carolina
  - Aventiv Research, Inc., Columbus, Ohio
  - Urologic Consultants of SE Pennsylvania, Bala-Cynwyd, Pennsylvania
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - University Diabetes Endocrine Consultants, Chattanooga, Tennessee
  - Centex Studies, Inc., Houston, Texas
  - Pioneer Research Solutions, Inc., Houston, Texas
  - Advanced Clinical Research, West Jordan, Utah
  - Clinical Research Associates of Tidewater, Norfolk, Virginia
  - National Clinical Research, Inc., Richmond, Virginia
  - Rainier Clinical Research Center, Inc., Renton, Washington
  - Mid-Columbia Research, Richland, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bernstein JS, Dhingra OP. A phase III, single-arm, 6-month trial of a wide-dose range oral testosterone undecanoate product. Ther Adv Urol. 2024 Apr 10;16:17562872241241864. doi: 10.1177/17562872241241864. eCollection 2024 Jan-Dec. PMID 38606384
- See also: MRS-TU-2019EXT study — https://clinicaltrials.gov/ct2/show/NCT04467697
- See also: Effects of Oral Testosterone Undecanoate (Kyzatrex) Versus Testosterone Gel (Androgel) on Long-Term (to 12 months) Blood Pressure Levels — http://online.liebertpub.com/doi/10.1089/andro.2022.0011

RESULTS

PARTICIPANT FLOW:
Groups:
- SOV2012-F1-Treated: 200 patients treated with SOV2012-F1, starting dose of 600 mg - (400 mg with morning meal and 200 mg with evening meal). Dose titrated (Days 28 and 56) up to a maximum of 600 mg TU in the morning and 400 mg in the evening or down to 200 mg TU in the morning based on plasma T at Days 14 and 42.
  SOV2012-F1: oral preparation of testosterone undecanoate (TU)
- Andro-Gel™ Treated: 100 patients treated with AndroGel, according to label, using samples on Days 14 and 42 with dose adjustment on Days 28 and 56.
  AndroGel: topical testosterone gel, 1.62%
Period: Overall Study
Arm/Group | SOV2012-F1-Treated | Andro-Gel™ Treated
Started | 214 | 100
Completed (Day 365. Five subjects withdrew from treatment or were lost to follow up after Day 365) | 162 | 76
Not Completed | 52 | 24
Not completed — Adverse Event | 10 | 5
Not completed — Lost to Follow-up | 21 | 7
Not completed — Physician Decision | 7 | 2
Not completed — Withdrawal by Subject | 14 | 10

BASELINE CHARACTERISTICS:
Population: Safety Set
Groups:
- Andro-Gel™ Treated: 100 patients treated with AndroGel, according to label, using sampling on Days 14 and 42 with dose adjustment on Days 28 and 56.
  AndroGel: topical testosterone gel, 1.62%
- Total: Total of all reporting groups
Arm/Group | SOV2012-F1-Treated | Andro-Gel™ Treated | Total
Number analyzed (Participants) | 214 | 100 | 314
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (9.15) | 50.7 (9.30) | 49.7 (9.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 214 | 100 | 314
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 55 | 27 | 82
  Not Hispanic or Latino | 159 | 73 | 232
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 34 | 11 | 45
  White | 171 | 86 | 257
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 1 | 8
Weight at Baseline [Mean (Standard Deviation); unit: kg] | 108.48 (22.827) | 108.97 (24.544) | 108.63 (23.349)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 34.12 (7.056) | 34.33 (6.486) | 34.19 (6.870)
Assigned breakfast diet [Count of Participants; unit: Participants] — Population: Data not collected for participants in the Androgel Treated Arm
  Participants
    Low-fat Breakfast: number analyzed (Participants) | 214 | 0 | 214
    Low-fat Breakfast | 27 |  | 27
    Normal-fat Breakfast: number analyzed (Participants) | 214 | 0 | 214
    Normal-fat Breakfast | 54 |  | 54
    High-fat Breakfast: number analyzed (Participants) | 214 | 0 | 214
    High-fat Breakfast | 130 |  | 130
    Missing: number analyzed (Participants) | 214 | 0 | 214
    Missing | 3 |  | 3
Diabetic Status [Count of Participants; unit: Participants]
  With Diabetes Mellitus | 31 | 13 | 44
  Without Diabetes Mellitus | 183 | 87 | 270
Hypertensive Status [Count of Participants; unit: Participants]
  Hypertensive | 127 | 60 | 187
  Not Hypertensive | 87 | 40 | 127
Hypertensive Treatment Status [Count of Participants; unit: Participants]
  With Antihypertensive Therapy at Visit 3 (Day 1) | 67 | 43 | 110
  Without Antihypertensive Therapy at Visit 3 (Day 1) | 147 | 57 | 204
Hypogonadal Status [Count of Participants; unit: Participants]
  Primary | 8 | 3 | 11
  Secondary | 206 | 97 | 303

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Male Hypogonadal Subjects With Average NaF/EDTA Plasma Total Testosterone (T Cavg) Within the Normal Range Using Oral SOV2012-F1.
Description: Efficacy assessment includes T Cavg calculated from NaF/EDTA plasma testosterone. The T Cavg is calculated as the 24-hour area under the curve (AUC), divided by 24, at Day 90, based on a fifteen blood samples (PK samples) taken over the 24-hours. The T concentration in each sample is measured using a validated LC-MS/MS method. The use of NaF/EDTA plasma tubes chilled after sample collection provides the most accurate values, as the prodrug TU may degrade post-sample collection, artificially inflating testosterone values.
Time Frame: 90 days
Population: Efficacy Set
Measure: Count of Participants; unit: Participants
Groups:
- SOV2012-F1 Treated: 200 patients treated with SOV2012-F1, starting dose of 600 mg - (400 mg with morning meal and 200 mg with evening meal). Dose titrated up to (Days 28 and 56) up to a maximum of 600 mg TU in the morning and 400 mg in the evening or down to 200 mg TU in the morning based on plasma T at Days 14 and 42.
  SOV2012-F1: oral preparation of testosterone undecanoate (TU)
Arm/Group | SOV2012-F1 Treated
Number analyzed (Participants) | 185
Participants | 166

2. Secondary Outcome: Percentages of Participants in Each Category for Maximum Plasma Concentration
Description: To determine the percentage of treated subjects with maximum plasma testosterone concentration (T Cmax) values (a) < 1.5X Upper Limit of Normal (ULN); (b) 1.8X to 2.5X ULN; and (c) > 2.5X ULN. For NaF/EDTA plasma, thresholds are 1200, 1440 and 2000 ng/dL of T. For serum, thresholds are 1500, 1800 and 2500 ng/dL of T. Note that the endpoint concerns only the investigational treatment SOV2012-F1 and the AndroGel results are reported for completeness. The reported percentages do not sum to 100% as the FDA criteria do not specify the percentage of subjects in the window of ≥ 1.5X and ≤ 1.8X the ULN.
Time Frame: 90 days
Population: Full Analysis Set
Measure: Number; unit: percentage of actual number of subjects
Groups:
- SOV2012-F1 Treated: 200 patients treated with SOV2012-F1, starting dose of 600 mg - (400 mg with morning meal and 200 mg with evening meal). Dose titrated (Days 28 and 56) up to a maximum of 600 mg TU in the morning and 400 mg in the evening or down to 200 mg TU in the morning based on plasma T at Days 14 and 42.
  SOV2012-F1: oral preparation of testosterone undecanoate (TU)
- Andro-gel™ Treated: 100 patients treated with AndroGel, according to label, using sampling on Days 14 and 42 with dose adjustment on Days 28 and 65.
  AndroGel: topical testosterone gel, 1.62%
Arm/Group | SOV2012-F1 Treated | Andro-gel™ Treated
Number analyzed (Participants) | 186 | 90
percentage of actual number of subjects
  T Cmax < 1200 ng/dL for SOV2012-F1; T Cmax < 1500 ng/dL for Andro-gel after 90 days | 76.9 | 92.2
  T Cmax 1440 to 2000 ng/dL for SOV2012-F1; T Cmax 1800 to 2500 ng/dL for Andro-gel after 90 days | 7.5 | 2.2
  T Cmax > 2000 ng/dL for SOV2012-F1; T Cmax > 2500 ng/dL for Andro-gel after 90days | 3.2 | 1.1

3. Other Pre Specified Outcome: Change From Baseline in the IPSS
Description: Patient reported outcomes will be assessed by the International Prostate Symptom Score (I-PSS) Reporting a score on a scale 0 to 35 (asymptomatic to very symptomatic). Mean change from baseline is reported and is the difference between the score at Baseline (pre-treatment) and at Day 90 and Day 365. Thus, a positive value at Day 90 or Day 365 represents an increase in the score from baseline.
Time Frame: Baseline (pre-treatment) to 90 days and 365 days
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SOV2012-F1 Treated | Andro-gel™ Treated
Number analyzed (Participants) | 214 | 100
score on a scale
  Baseline: number analyzed (Participants) | 211 | 100
  Baseline | 4.4 (4.12) | 5.4 (4.94)
  Change from baseline (Visit 8 - Day 90): number analyzed (Participants) | 184 | 90
  Change from baseline (Visit 8 - Day 90) | 0.2 (3.56) | 0.7 (3.72)
  Change from baseline (Visit Day 365): number analyzed (Participants) | 152 | 76
  Change from baseline (Visit Day 365) | 0.6 (3.99) | 1.0 (3.73)

4. Other Pre Specified Outcome: Change From Baseline in the Psychosexual Daily Questionnaire (PDQ)
Description: Patient reported outcomes are 7-day average score at baseline, and average change from baseline (CfB) at Day 90 and Day 365. Weekly daily average scores calculated for diaries completed at least 3 of 7 days.
  The three domains are:
  Sexual desire subscale 0=None, 1=very low to 7=Very High. Sexual enjoyment with/without partner subscale 0=None to 7=Very high enjoyment/pleasure. Partner availability not used in scoring. Positive CfB desirable.
  Positive and negative mood subscales 0=Not at all true to 7=Very true (Likert 7-point scale, 7-day average reported). Positive mood (sum of 4 questions) score range = 0 to 28; positive changes from baseline desirable. Negative mood (sum of 5 questions) score range = 0 to 35; negative CfB desirable.
  Weekly sexual activity subscale score is 7*(# of activities per week / # of days reported). Percent full erection uses scale of 0-100% (10% steps). Satisfaction with erection 0=not satisfactory to 7=very satisfactory. Positive CfB desirable.
Time Frame: Baseline (pre-treatment) to 90 days and 365 days
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SOV2012-F1 Treated | Andro-gel™ Treated
Number analyzed (Participants) | 214 | 100
score on a scale
  Overall Level of sexual desire Visit 3 - Day 1 (baseline): number analyzed (Participants) | 153 | 74
  Overall Level of sexual desire Visit 3 - Day 1 (baseline) | 1.990 (1.4195) | 2.039 (1.5659)
  Overall Level of sexual desire Visit 8 - Day 90: number analyzed (Participants) | 138 | 72
  Overall Level of sexual desire Visit 8 - Day 90 | 1.674 (1.6851) | 1.256 (1.5583)
  Overall Level of sexual desire Visit Day 365: number analyzed (Participants) | 144 | 68
  Overall Level of sexual desire Visit Day 365 | 1.552 (1.7596) | 1.372 (1.6968)
  Without a Partner Visit 3 - Day 1 (baseline): number analyzed (Participants) | 151 | 74
  Without a Partner Visit 3 - Day 1 (baseline) | 0.754 (0.9640) | 0.875 (1.1397)
  Without a Partner Visit 8 - Day 90: number analyzed (Participants) | 137 | 72
  Without a Partner Visit 8 - Day 90 | 0.742 (1.6478) | 0.498 (1.2075)
  Without a Partner Visit Day 365: number analyzed (Participants) | 143 | 68
  Without a Partner Visit Day 365 | 0.920 (1.5566) | 0.769 (1.5840)
  With a Partner Visit 3 - Day 1 (baseline): number analyzed (Participants) | 150 | 74
  With a Partner Visit 3 - Day 1 (baseline) | 0.954 (1.2033) | 0.840 (1.2928)
  With a Partner Visit 8 - Day 90: number analyzed (Participants) | 137 | 72
  With a Partner Visit 8 - Day 90 | 1.168 (1.7335) | 0.594 (1.7373)
  With a Partner Visit Day 365: number analyzed (Participants) | 142 | 66
  With a Partner Visit Day 365 | 1.106 (1.6670) | 0.760 (1.8284)
  Negative Mood Visit 3 - Day 1 (baseline): number analyzed (Participants) | 152 | 74
  Negative Mood Visit 3 - Day 1 (baseline) | 9.258 (5.8557) | 9.847 (5.0938)
  Negative Mood Visit 8 - Day 90: number analyzed (Participants) | 138 | 72
  Negative Mood Visit 8 - Day 90 | -2.205 (5.6199) | -1.886 (5.5670)
  Negative Mood Visit Day 365: number analyzed (Participants) | 144 | 68
  Negative Mood Visit Day 365 | -3.011 (5.3399) | -1.435 (5.7065)
  Positive mood - Visit 3 - Day 1 (baseline): number analyzed (Participants) | 152 | 74
  Positive mood - Visit 3 - Day 1 (baseline) | 16.799 (5.1778) | 15.742 (5.5015)
  Positive mood - Visit 8 - Day 90: number analyzed (Participants) | 138 | 72
  Positive mood - Visit 8 - Day 90 | 2.513 (5.0149) | 3.347 (5.2716)
  Positive mood - Day 365: number analyzed (Participants) | 144 | 68
  Positive mood - Day 365 | 3.407 (5.1065) | 2.817 (5.1714)
  Sexual Activity Score Visit 3 - Day 1 (baseline): number analyzed (Participants) | 152 | 74
  Sexual Activity Score Visit 3 - Day 1 (baseline) | 15.314 (13.8521) | 12.581 (12.0706)
  Sexual Activity Score Visit 8 - Day 90: number analyzed (Participants) | 138 | 72
  Sexual Activity Score Visit 8 - Day 90 | 12.284 (15.9338) | 10.951 (17.4041)
  Sexual Activity Score Day 365: number analyzed (Participants) | 144 | 68
  Sexual Activity Score Day 365 | 12.009 (16.5438) | 12.591 (17.7272)
  Erection Grade, Visit 3 - Day 1 (baseline): number analyzed (Participants) | 114 | 46
  Erection Grade, Visit 3 - Day 1 (baseline) | 32.145 (22.9941) | 30.652 (23.9078)
  Erection Grade, Visit 8 - Day 90: number analyzed (Participants) | 101 | 42
  Erection Grade, Visit 8 - Day 90 | 17.494 (25.0678) | 12.619 (22.6952)
  Erection Grade, Day 365: number analyzed (Participants) | 96 | 38
  Erection Grade, Day 365 | 14.235 (28.9806) | 17.584 (23.1670)
  Erection Duration, Visit 3 - Day 1 (baseline): number analyzed (Participants) | 114 | 46
  Erection Duration, Visit 3 - Day 1 (baseline) | 1.985 (1.4894) | 1.814 (1.5321)
  Erection Duration, Visit 8 - Day 90: number analyzed (Participants) | 101 | 42
  Erection Duration, Visit 8 - Day 90 | 1.480 (1.7137) | 1.012 (1.7166)
  Erection Duration, Day 365: number analyzed (Participants) | 95 | 38
  Erection Duration, Day 365 | 1.300 (1.8420) | 1.501 (1.6751)

5. Other Pre Specified Outcome: Change From Baseline in the SF-36
Description: Patient reported outcomes assessed by the Short-Form Survey (SF-36). This scale assesses 8 health concepts:
  1. limitations in physical activities because of health problems
  2. limitations in social activities because of physical or emotional problems
  3. limitations in usual role activities because of physical health problems
  4. bodily pain
  5. general mental health (psychological distress and well-being)
  6. limitations in usual role activities because of emotional problems
  7. vitality (energy and fatigue)
  8. general health perceptions.
  Each domain is scored from 0-100 with a score of 0 = maximum disability and a score of 100 = no disability.
  End of Treatment (EOT) occurred either at time of early withdrawal from the study or at Day 365. The reported value is the change from baseline. A positive value at EOT indicates improvement in the measure towards less disability. The EOT Change from Baseline is simply the arithmetic difference between the Baseline and EOT scores.
Time Frame: Baseline (Day 1, pre-treatment) and change from baseline at the End of Treatment (EOT)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SOV2012-F1-Treated | Andro-Gel™ Treated
Number analyzed (Participants) | 214 | 100
score on a scale
  Emotional Well-being (Baseline): number analyzed (Participants) | 190 | 90
  Emotional Well-being (Baseline) | 72.4 (17.55) | 68.0 (18.98)
  Emotional Well-being (End of Treatment): number analyzed (Participants) | 149 | 75
  Emotional Well-being (End of Treatment) | 7.1 (15.44) | 5.6 (15.37)
  Energy/Fatigue (Baseline): number analyzed (Participants) | 168 | 83
  Energy/Fatigue (Baseline) | 61.0 (20.22) | 53.0 (21.91)
  Energy/Fatigue (End of Treatment): number analyzed (Participants) | 149 | 75
  Energy/Fatigue (End of Treatment) | 16.6 (21.00) | 15.5 (21.12)
  General Health (Baseline): number analyzed (Participants) | 168 | 83
  General Health (Baseline) | 69.0 (17.09) | 67.0 (18.33)
  General Health (End of Treatment): number analyzed (Participants) | 149 | 75
  General Health (End of Treatment) | 3.5 (16.87) | 6.9 (15.46)
  Health Change (Baseline): number analyzed (Participants) | 168 | 83
  Health Change (Baseline) | 65.2 (20.66) | 59.6 (18.66)
  Health Change (End of Treatment): number analyzed (Participants) | 149 | 75
  Health Change (End of Treatment) | 14.6 (26.81) | 7.0 (24.16)
  Pain (Baseline): number analyzed (Participants) | 168 | 83
  Pain (Baseline) | 77.17 (21.103) | 70.57 (22.619)
  Pain (End of Treatment): number analyzed (Participants) | 148 | 75
  Pain (End of Treatment) | 4.16 (21,778) | 1.43 (21.834)
  Physical Functioning (Baseline): number analyzed (Participants) | 168 | 83
  Physical Functioning (Baseline) | 85.5 (19.03) | 83.3 (19.05)
  Physical Functioning (End of Treatment): number analyzed (Participants) | 149 | 75
  Physical Functioning (End of Treatment) | 3.6 (17.57) | 6.8 (19.82)
  Role Limitations due to Emotional Problems (Baseline): number analyzed (Participants) | 168 | 83
  Role Limitations due to Emotional Problems (Baseline) | 85.317 (30.2358) | 79.116 (34.4177)
  Role Limitations due to Emotional Problems (End of Treatment): number analyzed (Participants) | 149 | 75
  Role Limitations due to Emotional Problems (End of Treatment) | 12.081 (39.3671) | 5.778 (35.2483)
  Role Limitations due to Physical Health (Baseline): number analyzed (Participants) | 168 | 83
  Role Limitations due to Physical Health (Baseline) | 82.1 (31.09) | 75.0 (35.14)
  Role Limitations due to Physical Health (End of Treatment): number analyzed (Participants) | 149 | 75
  Role Limitations due to Physical Health (End of Treatment) | 12.4 (41.06) | 14.3 (39.67)
  Social Functioning (Baseline): number analyzed (Participants) | 168 | 83
  Social Functioning (Baseline) | 84.75 (18.527) | 83.73 (18.799)
  Social Functioning (End of Treatment): number analyzed (Participants) | 149 | 75
  Social Functioning (End of Treatment) | 9.31 (22.140) | 6.83 (22.161)
  Mental Health Composite (Baseline): number analyzed (Participants) | 168 | 83
  Mental Health Composite (Baseline) | 51.885 (8.6492) | 49.025 (10.5313)
  Mental Health Composite (End of Treatment): number analyzed (Participants) | 149 | 75
  Mental Health Composite (End of Treatment) | 5.478 (9.8093) | 3.515 (9.1373)
  Physical Health Composite (Baseline): number analyzed (Participants) | 168 | 83
  Physical Health Composite (Baseline) | 49.229 (8.3286) | 48.002 (8.7737)
  Physical Health Composite (End of Treatment): number analyzed (Participants) | 149 | 75
  Physical Health Composite (End of Treatment) | 1.558 (7.5381) | 2.968 (8.1428)

6. Other Pre Specified Outcome: Change From Baseline in the IIEF
Description: Patient reported outcomes are assessed by the International Index of Erectile Function (IIEF). A score of 0-5 (higher score indicating improvement) is awarded to each of the 15 questions that examine overall satisfaction (2 questions, total possible score=10), and the 4 main domains of male sexual function: erectile function (6 questions, total possible score=30), orgasmic function (2 questions, total possible score=10), sexual desire (2 questions, total possible score=10), and intercourse satisfaction (3 questions, total possible score=15).
  The IIEF results are reported at Baseline (Day 1, pre-treatment) and the change from baseline at the End of Treatment (EOT). EOT occurred either at time of early withdrawal from the study or at Day 365.
  The reported value is the change from baseline. A positive value at EOT indicates improvement in the measure. The EOT Change from Baseline is simply the arithmetic difference between the Baseline and End of Treatment scores.
Time Frame: Baseline (Day 1, pre-treatment) and change from baseline at the End of Treatment (EOT)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SOV2012-F1-Treated | Andro-Gel™ Treated
Number analyzed (Participants) | 214 | 100
score on a scale
  Erectile Function (Baseline): number analyzed (Participants) | 157 | 76
  Erectile Function (Baseline) | 19.8 (8.99) | 17.1 (9.62)
  Erectile Function (End of Treatment): number analyzed (Participants) | 157 | 76
  Erectile Function (End of Treatment) | 5.1 (8.30) | 4.1 (8.35)
  Intercourse Satisfaction (Baseline): number analyzed (Participants) | 157 | 76
  Intercourse Satisfaction (Baseline) | 8.4 (5.17) | 6.8 (5.55)
  Intercourse Satisfaction (End of Treatment): number analyzed (Participants) | 157 | 76
  Intercourse Satisfaction (End of Treatment) | 2.4 (4.56) | 2.4 (4.81)
  Orgasmic Function (Baseline): number analyzed (Participants) | 157 | 76
  Orgasmic Function (Baseline) | 7.3 (3.45) | 6.7 (3.42)
  Orgasmic Function (End of Treatment): number analyzed (Participants) | 157 | 76
  Orgasmic Function (End of Treatment) | 1.5 (3.61) | 2.4 (4.81)
  Sexual Desire (Baseline): number analyzed (Participants) | 157 | 76
  Sexual Desire (Baseline) | 3.6 (1.12) | 3.7 (1.10)
  Sexual Desire (End of Treatment): number analyzed (Participants) | 157 | 76
  Sexual Desire (End of Treatment) | 0.7 (1.25) | 0.9 (1.10)
  Overall Satisfaction (Baseline) | 4.8 (2.31) | 4.1 (2.27)
  Overall Satisfaction Visit Day 365 | 2.3 (2.55) | 1.6 (2.83)

7. Other Pre Specified Outcome: Change From Baseline in Fasting Serum Glucose (FSG) Concentration
Description: The measured value is the FSG concentration reported as mg/dL. The FSG results are reported at Baseline (Day 1, pre-treatment) and the change from baseline at Day 90, Day 180, Day 270 and the End of Treatment. End of treatment occurred either at time of early withdrawal from the study or at Day 365.
  The reported value is the change from baseline. The Change from Baseline is simply the arithmetic difference between the Baseline and measured values.
Time Frame: Baseline (Day 1, pre-treatment) and the change from baseline at Day 90, Day 180, Day 270 and the End of Treatment.
Population: Safety Set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | SOV2012-F1-Treated | Andro-Gel™ Treated
Number analyzed (Participants) | 214 | 100
mg/dL
  Baseline: number analyzed (Participants) | 213 | 100
  Baseline | 108.6 (31.19) | 110.3 (26.01)
  Visit 8 - Day 90: number analyzed (Participants) | 183 | 87
  Visit 8 - Day 90 | 4.2 (24.84) | 3.0 (23.51)
  Visit 10 - Day 180: number analyzed (Participants) | 169 | 82
  Visit 10 - Day 180 | 1.4 (24.54) | 2.4 (21.48)
  Visit 12 - Day 270: number analyzed (Participants) | 164 | 77
  Visit 12 - Day 270 | 1.4 (21.82) | 6.2 (31.97)
  End of Treatment: number analyzed (Participants) | 154 | 71
  End of Treatment | -4.7 (20.41) | -0.8 (21.61)

8. Other Pre Specified Outcome: Change From Baseline in Fasting Insulin Concentration
Description: The measured value is the insulin concentration reported as in units of uU/mL. The insulin results are reported at Baseline (Day 1, pre-treatment) and the change from baseline at Day 90, Day 180, Day 270 and the End of Treatment. End of treatment occurred either at time of early withdrawal from the study or at Day 365.
  The reported value is the change from baseline. The Change from Baseline is simply the arithmetic difference between the Baseline and measured values.
Time Frame: Baseline (Day 1, pre-treatment) and the change from baseline at Day 90, Day 180, Day 270 and the End of Treatment.
Population: Safety Set
Measure: Mean (Standard Deviation); unit: uU/mL
Arm/Group | SOV2012-F1-Treated | Andro-Gel™ Treated
Number analyzed (Participants) | 214 | 100
uU/mL
  Baseline: number analyzed (Participants) | 213 | 98
  Baseline | 27.30 (38.030) | 24.83 (18.555)
  Visit 8 - Day 90: number analyzed (Participants) | 187 | 87
  Visit 8 - Day 90 | 3.59 (56.110) | 2.43 (19.328)
  Visit 10 - Day 180: number analyzed (Participants) | 172 | 80
  Visit 10 - Day 180 | 2.77 (54.045) | 5.12 (46.035)
  Visit 12 - Day 270: number analyzed (Participants) | 165 | 75
  Visit 12 - Day 270 | 5.12 (63.889) | 0.54 (20.026)
  End of Treatment: number analyzed (Participants) | 153 | 71
  End of Treatment | -5.24 (43.047) | -2.58 (14.967)

9. Other Pre Specified Outcome: Change From Baseline in Blood Pressures After Oral Testosterone Undecanoate and Testosterone Gel
Description: Changes from baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP), as mmHg.
  The blood pressure results are reported at Baseline (Day 1, pre-treatment) and the change from baseline at Day 90, Day 180, Day 270 and the End of Treatment. End of treatment occurred either at time of early withdrawal from the study or at Day 365.
  The reported value is the change from baseline. The Change from Baseline is simply the arithmetic difference between the Baseline and the measured value. A positive value for Change in Baseline represents an increase in the measured SBP or DBP.
Time Frame: Baseline (Day 1, pre-treatment) and the change from baseline at Day 90, Day 180, Day 270 and the End of Treatment.
Population: Safety Set
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SOV2012-F1-Treated | Andro-Gel™ Treated
Number analyzed (Participants) | 214 | 100
mmHg
  Clinic systolic BP - Baseline | 125.8 (9.122) | 125.95 (10.130)
  Clinic systolic BP - 90 day: number analyzed (Participants) | 180 | 89
  Clinic systolic BP - 90 day | 2.16 (10.400) | 3.07 (9.797)
  Clinic systolic BP - 180 day: number analyzed (Participants) | 161 | 79
  Clinic systolic BP - 180 day | 1.89 (10.174) | 1.91 (9.044)
  Clinic systolic BP - 365 day: number analyzed (Participants) | 136 | 70
  Clinic systolic BP - 365 day | 2.75 (9.501) | 3.38 (10.492)
  Clinic diastolic BP - Baseline | 78.88 (6.340) | 79.19 (6.624)
  Clinic diastolic BP - 90 day: number analyzed (Participants) | 180 | 89
  Clinic diastolic BP - 90 day | 0.58 (6.800) | 1.10 (8.262)
  Clinic diastolic BP - 180 day: number analyzed (Participants) | 161 | 79
  Clinic diastolic BP - 180 day | 0.67 (6.014) | 2.60 (6.826)
  Clinic diastolic BP - 365 day: number analyzed (Participants) | 136 | 70
  Clinic diastolic BP - 365 day | 1.14 (6.119) | 1.75 (7.213)

10. Other Pre Specified Outcome: Change From Baseline in Liver Function Tests
Description: Liver function tests (ALT, AST, total bilirubin, alkaline phosphatase). The liver function test results are reported at Baseline (Day 1, pre-treatment) and the change from baseline at Day 90, Day 180, Day 270 and the End of Treatment. End of treatment occurred either at time of early withdrawal from the study or at Day 365.
  The reported value is the change from baseline. The Change from Baseline is simply the arithmetic difference between the Baseline and the measured value. A positive value for Change in Baseline represents an increase in the liver function test value
Time Frame: Baseline (Day 1, pre-treatment) and the change from baseline at Day 90, Day 180, Day 270 and the End of Treatment.
Population: Safety set
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | SOV2012-F1-Treated | Andro-Gel™ Treated
Number analyzed (Participants) | 214 | 100
U/L
  Alkaline Phosphatase (Baseline) | 72.8 (18.79) | 74.0 (20.19)
  Alkaline Phosphatase (Visit 8 - Day 90): number analyzed (Participants) | 183 | 87
  Alkaline Phosphatase (Visit 8 - Day 90) | -6.0 (11.03) | -1.2 (8.90)
  Alkaline Phosphatase (Visit 10 - Day 180): number analyzed (Participants) | 170 | 82
  Alkaline Phosphatase (Visit 10 - Day 180) | -4.2 (12.14) | -1.6 (10.13)
  Alkaline Phosphatase (Visit 12 - Day 270): number analyzed (Participants) | 165 | 77
  Alkaline Phosphatase (Visit 12 - Day 270) | -5.5 (10.57) | -2.1 (9.96)
  Alkaline Phosphatase (Visit Day 365): number analyzed (Participants) | 157 | 75
  Alkaline Phosphatase (Visit Day 365) | -4.5 (11.42) | -1.5 (10.38)
  Alkaline Phosphatase (End of Treatment): number analyzed (Participants) | 180 | 89
  Alkaline Phosphatase (End of Treatment) | -4.0 (11.31) | -1.5 (10.37)
  Alanine Aminotransferase (ALT) - Baseline | 30.5 (13.59) | 31.0 (12.64)
  Alanine Aminotransferase (ALT), Visit 8 - Day 90: number analyzed (Participants) | 182 | 87
  Alanine Aminotransferase (ALT), Visit 8 - Day 90 | -2.6 (14.28) | -0.0 (13.30)
  Alanine Aminotransferase (ALT), Visit 10 - Day 180: number analyzed (Participants) | 170 | 81
  Alanine Aminotransferase (ALT), Visit 10 - Day 180 | -2.9 (11.44) | 0.9 (16.64)
  Alanine Aminotransferase (ALT), Visit 12 - Day 270: number analyzed (Participants) | 165 | 77
  Alanine Aminotransferase (ALT), Visit 12 - Day 270 | -2.2 (12.76) | 0.7 (17.25)
  Alanine Aminotransferase (ALT), Visit Day 365: number analyzed (Participants) | 157 | 75
  Alanine Aminotransferase (ALT), Visit Day 365 | -1.4 (12.89) | 1.3 (14.55)
  Alanine Aminotransferase (ALT) - End of Treatment: number analyzed (Participants) | 180 | 89
  Alanine Aminotransferase (ALT) - End of Treatment | -0.4 (19.84) | 0.9 (14.64)
  Aspartate Aminotransferase (AST) - Baseline | 23.8 (8.83) | 23.4 (8.04)
  Aspartate Aminotransferase (AST) - Visit 8, Day 90: number analyzed (Participants) | 182 | 87
  Aspartate Aminotransferase (AST) - Visit 8, Day 90 | 0.8 (10.96) | 1.2 (8.34)
  Aspartate Aminotransferase (AST) - Visit 10, Day 180: number analyzed (Participants) | 170 | 82
  Aspartate Aminotransferase (AST) - Visit 10, Day 180 | 0.1 (8.04) | 1.7 (12.24)
  Aspartate Aminotransferase (AST) - Visit 12, Day 270: number analyzed (Participants) | 165 | 77
  Aspartate Aminotransferase (AST) - Visit 12, Day 270 | 0.0 (9.03) | 0.3 (11.27)
  Aspartate Aminotransferase (AST) - Visit Day 365: number analyzed (Participants) | 157 | 75
  Aspartate Aminotransferase (AST) - Visit Day 365 | 2.2 (27.18) | 1.2 (9.64)
  Aspartate Aminotransferase (AST) - End of Treatment: number analyzed (Participants) | 180 | 89
  Aspartate Aminotransferase (AST) - End of Treatment | 2.4 (27.18) | 1.0 (9.69)

11. Other Pre Specified Outcome: Change in Bilirubin
Description: Change in bilirubin from Baseline The bilirubin test results are reported at Baseline (Day 1, pre-treatment) and the change from baseline at Day 90, Day 180, Day 270 and the End of Treatment. End of treatment occurred either at time of early withdrawal from the study or at Day 365.
  The reported value is the change from baseline. The Change from Baseline is simply the arithmetic difference between the Baseline and the measured value. A positive value for Change in Baseline represents an increase in the bilirubin value.
Time Frame: Baseline (Day 1, pre-treatment) and the change from baseline at Day 90, Day 180, Day 270 and the End of Treatment.
Population: Safety set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | SOV2012-F1-Treated | Andro-Gel™ Treated
Number analyzed (Participants) | 214 | 100
mg/dL
  Bilirubin - Baseline | 0.491 (0.2437) | 0.465 (0.2561)
  Bilirubin, Visit 8 - Day 90: number analyzed (Participants) | 182 | 87
  Bilirubin, Visit 8 - Day 90 | -0.088 (0.2024) | -0.058 (0.2231)
  Bilirubin, Visit 10 - Day 180: number analyzed (Participants) | 170 | 82
  Bilirubin, Visit 10 - Day 180 | -0.007 (0.2350) | -0.004 (0.2106)
  Bilirubin, Visit 12 - Day 270: number analyzed (Participants) | 165 | 77
  Bilirubin, Visit 12 - Day 270 | 0.013 (0.2254) | 0.029 (0.2171)
  Bilirubin, Visit Day 365: number analyzed (Participants) | 157 | 75
  Bilirubin, Visit Day 365 | -0.027 (0.2155) | 0.038 (0.2245)
  Bilirubin, End of Treatment: number analyzed (Participants) | 180 | 89
  Bilirubin, End of Treatment | -0.032 (0.2157) | 0.026 (0.2117)

12. Other Pre Specified Outcome: Change From Baseline in Hematology Parameters
Description: Hematology parameters (HbA1c) with diabetes mellitus and Without diabetes mellitus.
  The HbA1c test results are reported at Baseline (Day 1, pre-treatment) and the change from baseline at the End of Treatment. End of treatment occurred either at time of early withdrawal from the study or at Day 365.
  The reported value at End of Treatment is the change from baseline. The Change from Baseline is simply the arithmetic difference between the Baseline and the End of Treatment value. Normal range for HbA1c is 4 to 5.6%, pre-diabetic is 5.7 to 6.4%, and diabetic is equal to or greater than 6.5%.
Time Frame: Baseline (Day 1, pre-treatment) and the change from baseline at the End of Treatment
Population: Safety Set
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | SOV2012-F1-Treated | Andro-Gel™ Treated
Number analyzed (Participants) | 214 | 100
percentage of HbA1c
  HbA1c with diabetes mellitus (baseline): number analyzed (Participants) | 31 | 13
  HbA1c with diabetes mellitus (baseline) | 7.20 (0.515) | 7.07 (0.340)
  HbA1c with diabetes mellitus end of treatment: number analyzed (Participants) | 27 | 12
  HbA1c with diabetes mellitus end of treatment | 0.04 (0.975) | 0.73 (0.608)
  HbA1c without diabetes mellitus (baseline): number analyzed (Participants) | 183 | 87
  HbA1c without diabetes mellitus (baseline) | 5.63 (0.432) | 5.65 (0.469)
  HbA1c without diabetes mellitus end of treatment: number analyzed (Participants) | 129 | 65
  HbA1c without diabetes mellitus end of treatment | 0.11 (0.369) | 0.00 (0.326)

13. Other Pre Specified Outcome: Change From Baseline in Hormone Levels
Description: Hormone levels (luteinizing hormone [LH], follicle-stimulating hormone [FSH], sex hormone-binding globulin [SHBG], TSH).
  The hormone level test results are reported at Baseline (Day 1, pre-treatment) and the change from baseline at Day 90, and the End of Treatment. End of treatment occurred either at time of early withdrawal from the study or at Day 365.
  The Change from Baseline is simply the arithmetic difference between the Baseline and the measured value at Day 90 or Day 365. A positive value for Change in Baseline represents an increase in the hormone level.
Time Frame: Baseline (Day 1, pre-treatment) and the change from baseline at Day 90, and the End of Treatment
Population: Safety set
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | SOV2012-F1-Treated | Andro-Gel™ Treated
Number analyzed (Participants) | 214 | 100
mIU/mL
  Follicle Stimulating Hormone (FSH) - Baseline | 5.46 (5.496) | 5.03 (3.283)
  Follicle Stimulating Hormone (FSH) - Visit 8 - Day 90: number analyzed (Participants) | 187 | 89
  Follicle Stimulating Hormone (FSH) - Visit 8 - Day 90 | -3.35 (4.423) | -3.28 (2.888)
  Follicle Stimulating Hormone (FSH) - Visit Day 365: number analyzed (Participants) | 157 | 76
  Follicle Stimulating Hormone (FSH) - Visit Day 365 | -2.72 (4.209) | -1.82 (6.708)
  Follicle Stimulating Hormone (FSH) - Visit Day 365 End of Treatment: number analyzed (Participants) | 180 | 89
  Follicle Stimulating Hormone (FSH) - Visit Day 365 End of Treatment | -2.45 (4.162) | -1.77 (6.230)
  Luteinizing Hormone (LH) - Baseline | 4.82 (3.755) | 4.58 (2.494)
  Luteinizing Hormone (LH) - Visit 8 - Day 90: number analyzed (Participants) | 187 | 89
  Luteinizing Hormone (LH) - Visit 8 - Day 90 | -3.25 (3.805) | -3.28 (2.472)
  Luteinizing Hormone (LH) - Visit Day 365: number analyzed (Participants) | 157 | 76
  Luteinizing Hormone (LH) - Visit Day 365 | -2.53 (3.487) | -1.67 (4.484)
  Luteinizing Visit Day Hormone (LH) - End of Treatment: number analyzed (Participants) | 180 | 89
  Luteinizing Visit Day Hormone (LH) - End of Treatment | -2.18 (3.582) | -1.60 (4.272)

14. Other Pre Specified Outcome: Change in Hormone SHBG
Description: Change in hormone Sex Hormone Binding Globulin (SHBG). The hormone level test results are reported at Baseline (Day 1, pre-treatment) and the change from baseline at Day 90, and the End of Treatment. End of treatment occurred either at time of early withdrawal from the study or at Day 365.
  The Change from Baseline is simply the arithmetic difference between the Baseline and the measured value at Day 90 or Day 365. A positive value for Change in Baseline represents an increase in the hormone level.
Time Frame: Baseline (Day 1, pre-treatment) and the change from baseline at Day 90, and the End of Treatment
Population: Safety Set
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | SOV2012-F1-Treated | Andro-Gel™ Treated
Number analyzed (Participants) | 214 | 100
nmol/L
  SHBG - Baseline: number analyzed (Participants) | 214 | 99
  SHBG - Baseline | 27.08 (11.958) | 24.52 (10.210)
  SHBG - Day 90: number analyzed (Participants) | 187 | 89
  SHBG - Day 90 | -8.99 (8.167) | 0.26 (4.341)
  SHBG - Day 365: number analyzed (Participants) | 156 | 73
  SHBG - Day 365 | -7.00 (9.326) | 1.60 (8.126)
  SHBG - End of Treatment: number analyzed (Participants) | 177 | 87
  SHBG - End of Treatment | -6.25 (9.637) | 1.39 (7.595)

15. Other Pre Specified Outcome: Change in TSH (Thyrotropin)
Description: Change from Baseline in Thyroid stimulating Hormone (TSH). The TSH test results are reported at Baseline (Day 1, pre-treatment) and the change from baseline at Day 90, and the End of Treatment. End of treatment occurred either at time of early withdrawal from the study or at Day 365.
  The Change from Baseline is simply the arithmetic difference between the Baseline and the measured value at Day 90 or Day 365. A positive value for Change in Baseline represents an increase in the TSH level.
Time Frame: Baseline (Day 1, pre-treatment) and the change from baseline at Day 90, and the End of Treatment
Population: Safety Set
Measure: Mean (Standard Deviation); unit: mU/L
Arm/Group | SOV2012-F1-Treated | Andro-Gel™ Treated
Number analyzed (Participants) | 214 | 100
mU/L
  Thyrotropin - Baseline | 2.212 (1.1941) | 2.407 (1.2624)
  Thyrotropin - Day 90: number analyzed (Participants) | 186 | 90
  Thyrotropin - Day 90 | 0.293 (1.0140) | 0.343 (1.0773)
  Thyrotropin - Day 365: number analyzed (Participants) | 157 | 76
  Thyrotropin - Day 365 | 0.195 (1.1494) | 0.122 (1.0080)
  Thyrotropin - End of Treatment: number analyzed (Participants) | 180 | 88
  Thyrotropin - End of Treatment | 0.209 (1.1204) | 0.081 (1.0571)

16. Other Pre Specified Outcome: Change From Baseline in Lipid Profiles
Description: Lipid profiles (high and low-density lipoproteins, total cholesterol, triglycerides).
  The lipid test results are reported at Baseline (Day 1, pre-treatment) and the change from baseline at Day 90, Day 180, Day 270, Day 365 and the End of Treatment. End of Treatment occurred either at time of early withdrawal from the study or at Day 365.
  The Change from Baseline is simply the arithmetic difference between the Baseline and the measured value. A positive value for Change in Baseline represents an increase in the lipid value.
Time Frame: Baseline (Day 1, pre-treatment) and the change from baseline at Day 90, Day 180, Day 270, Day 365 and the End of Treatment
Population: Safety Set LDL Cholesterol, Baseline = number of subjects with non-missing results
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | SOV2012-F1-Treated | Andro-Gel™ Treated
Number analyzed (Participants) | 214 | 100
mg/dL
  Cholesterol, Baseline | 190.5 (38.55) | 191.1 (39.12)
  Cholesterol, Visit 8 Day 90: number analyzed (Participants) | 184 | 88
  Cholesterol, Visit 8 Day 90 | -8.6 (29.86) | -6.1 (26.36)
  Cholesterol, Visit 10 Day 180: number analyzed (Participants) | 171 | 82
  Cholesterol, Visit 10 Day 180 | -10.7 (29.56) | -5.7 (25.07)
  Cholesterol, Visit 12 Day 270: number analyzed (Participants) | 165 | 77
  Cholesterol, Visit 12 Day 270 | -14.3 (32.28) | -8.2 (31.83)
  Cholesterol, Visit Day 365: number analyzed (Participants) | 157 | 75
  Cholesterol, Visit Day 365 | -14.0 (28.72) | -5.5 (38.41)
  Cholesterol, End of Treatment: number analyzed (Participants) | 180 | 89
  Cholesterol, End of Treatment | -11.6 (30.56) | -6.0 (36.24)
  HDL Cholesterol, Baseline | 46.8 (11.84) | 45.2 (11.33)
  HDL Cholesterol, Visit 8, Day 90: number analyzed (Participants) | 184 | 88
  HDL Cholesterol, Visit 8, Day 90 | -7.5 (8.45) | -1.5 (6.79)
  HDL Cholesterol, Visit 10, Day 180: number analyzed (Participants) | 171 | 82
  HDL Cholesterol, Visit 10, Day 180 | -6.9 (9.96) | -1.9 (6.94)
  HDL Cholesterol, Visit 12, Day 270: number analyzed (Participants) | 165 | 7
  HDL Cholesterol, Visit 12, Day 270 | -6.7 (9.53) | -1.6 (7.62)
  HDL Cholesterol, Visit Day 365: number analyzed (Participants) | 157 | 75
  HDL Cholesterol, Visit Day 365 | -7.9 (9.83) | -2.8 (7.12)
  HDL Cholesterol, End of Treatment: number analyzed (Participants) | 180 | 89
  HDL Cholesterol, End of Treatment | -7.1 (9.87) | -2.8 (7.05)
  LDL Cholesterol, Baseline 1: number analyzed (Participants) | 210 | 99
  LDL Cholesterol, Baseline 1 | 110.8 (34.72) | 108.9 (34.39)
  LDL Cholesterol, Visit 8 - Day 90: number analyzed (Participants) | 177 | 82
  LDL Cholesterol, Visit 8 - Day 90 | -0.3 (26.13) | -4.3 (22.91)
  LDL Cholesterol, Visit 10 - Day 180: number analyzed (Participants) | 165 | 73
  LDL Cholesterol, Visit 10 - Day 180 | -3.1 (25.79) | -5.4 (21.92)
  LDL Cholesterol, Visit 12 - Day 270: number analyzed (Participants) | 160 | 70
  LDL Cholesterol, Visit 12 - Day 270 | -6.1 (27.90) | -5.4 (26.84)
  LDL Cholesterol, Visit Day 365: number analyzed (Participants) | 154 | 68
  LDL Cholesterol, Visit Day 365 | -4.8 (25.06) | -5.4 (30.42)
  LDL Cholesterol, End of Treatment: number analyzed (Participants) | 173 | 80
  LDL Cholesterol, End of Treatment | -3.8 (25.92) | -5.5 (29.41)
  Triglycerides, Baseline | 167.6 (86.30) | 184.6 (86.79)
  Triglycerides, Visit 8 - Day 90: number analyzed (Participants) | 184 | 88
  Triglycerides, Visit 8 - Day 90 | -2.5 (86.21) | 9.4 (100.18)
  Triglycerides, Visit 10 - Day 180: number analyzed (Participants) | 171 | 82
  Triglycerides, Visit 10 - Day 180 | -3.2 (75.75) | 19.0 (99.18)
  Triglycerides, Visit 12 - Day 270: number analyzed (Participants) | 165 | 77
  Triglycerides, Visit 12 - Day 270 | -8.0 (88.60) | 15.4 (126.56)
  Triglycerides, Visit Day 365: number analyzed (Participants) | 157 | 75
  Triglycerides, Visit Day 365 | -7.0 (73.84) | 26.0 (144.41)
  Triglycerides, End of Treatment: number analyzed (Participants) | 180 | 89
  Triglycerides, End of Treatment | -4.8 (77.97) | 25.9 (136.57)

17. Other Pre Specified Outcome: Change From Baseline in PSA
Description: Serum prostate-specific antigen (PSA). The PSA results are reported at Baseline (Day 1, pre-treatment) and the change from baseline at Day 90, Day 180, Day 270, Day 365 and the End of Treatment. End of Treatment occurred either at time of early withdrawal from the study or at Day 365.
  The reported value is the change from baseline. The Change from Baseline is simply the arithmetic difference between the Baseline and the measured value. A positive value for Change in Baseline represents an increase in the PSA value.
Time Frame: as for outcome 16
Population: Safety Set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SOV2012-F1-Treated | Andro-Gel™ Treated
Number analyzed (Participants) | 214 | 100
ng/mL
  Prostate Specific Antigen, Baseline | 0.87 (0.549) | 0.78 (0.506)
  Prostate Specific Antigen, Visit 8 - Day 90: number analyzed (Participants) | 186 | 90
  Prostate Specific Antigen, Visit 8 - Day 90 | 0.18 (0.452) | 0.18 (0.435)
  Prostate Specific Antigen, Visit 10 - Day 180: number analyzed (Participants) | 173 | 82
  Prostate Specific Antigen, Visit 10 - Day 180 | 0.20 (0.472) | 0.22 (0.533)
  Prostate Specific Antigen, Visit 12 - Day 270: number analyzed (Participants) | 165 | 77
  Prostate Specific Antigen, Visit 12 - Day 270 | 0.25 (0.586) | 0.29 (0.650)
  Prostate Specific Antigen, Visit Day 365: number analyzed (Participants) | 157 | 76
  Prostate Specific Antigen, Visit Day 365 | 0.23 (0.525) | 0.27 (0.756)
  Prostate Specific Antigen, End of Treatment: number analyzed (Participants) | 180 | 88
  Prostate Specific Antigen, End of Treatment | 0.23 (0.523) | 0.41 (1.688)

18. Other Pre Specified Outcome: Effect of SOV2012-F1 on Adrenal Cortical Function as Assessed by Measuring the Cortisol Response to Synthetic ACTH at Baseline in Subjects
Description: To determine the effect of SOV2012-F1 on adrenal cortical function as assessed by measuring the cortisol response to synthetic ACTH at baseline and after 52 weeks of treatment in a subset of SOV2012-F1 subjects. . The sample size was calculated based on a assumed common Standard Deviation of 93 nmol/L to yield a half-width of not more than 60 nmol/L; hence a sample size of 30 was targeted for the investigational (SOV2012-F1) arm, and 15 for the safety control arm (AndroGel).
Time Frame: 52 weeks
Population: ACTH Completers Set
Measure: Mean (Standard Deviation); unit: nmol/L
Groups:
- SOV2012-F1-Treated: The ACTH Substudy enrolled 29 patients out of 200 patients treated with SOV2012-F1, starting dose of 600 mg - (400 mg with morning meal and 200 mg with evening meal). Dose titrated (Days 28 and 56) up to a maximum of 600 mg TU in the morning and 400 mg in the evening or down to 200 mg TU in the morning based on plasma T at Days 14 and 42.
  SOV2012-F1: oral preparation of testosterone undecanoate (TU)
- Andro-Gel™ Treated: The ACTH Substudy enrolled 13 participants out of the 100 patients treated with AndroGel, according to label, using samples on Days 14 and 42 with dose adjustment on Days 28 and 56.
  AndroGel: topical testosterone gel, 1.62%
Arm/Group | SOV2012-F1-Treated | Andro-Gel™ Treated
Number analyzed (Participants) | 29 | 13
nmol/L
  Maximum Serum Cortisol (Day 1 - Baseline) | 23.75 (3.584) | 25.68 (2.373)
  Maximum Serum Cortisol (Day 365 - End of Study) | 25.22 (4.561) | 27.05 (3.267)

ADVERSE EVENTS:
Time Frame: 365 days
Groups:
- SOV2012-F1-Treated: 200 patients treated with SOV2012-F1, starting dose of 600 mg - (400 mg with morning meal and 200 mg with evening meal). Dose titrated up to a maximum of 600 mg TU in the morning and 400 mg in the evening or down to 200 mg TU in the morning based on plasma T at Days 14 and 42.
  SOV2012-F1: oral preparation of testosterone undecanoate (TU)
- Andro-Gel Treated: 100 patients treated with AndroGel, according to label, using samples on Days 14 and 42 with dose adjustment on Days 28 and 56.
  AndroGel: topical testosterone gel, 1.62%
Arm/Group | SOV2012-F1-Treated | Andro-Gel Treated
All-Cause Mortality (participants affected / at risk) | 1/214 | 0/100
Serious Adverse Events (participants affected / at risk) | 9/214 | 1/100
Other Adverse Events (participants affected / at risk) | 53/214 | 25/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOV2012-F1-Treated (N=214) | Andro-Gel Treated (N=100)
Acute Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Renal tubular acidosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Finger amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOV2012-F1-Treated (N=214) | Andro-Gel Treated (N=100)
Upper respiratory tract infection (Infections and infestations) | 15 (20) | 12 (16)
Influenza (Infections and infestations) | 10 (10) | 4 (4)
Viral upper respiratory tract infection (Infections and infestations) | 7 (10) | 5 (6)
Sinusitis (Infections and infestations) | 5 (5) | 4 (4)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2)
Acute sinusitis (Infections and infestations) | 1 (1) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2)
Blood pressure increased (Investigations) | 7 (9) | 3 (3)
Prostatic specific antigen increased (Investigations) | 5 (5) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (9) | 6 (7)
Back Pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (5)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 2 (2)
Constipation (Gastrointestinal disorders) | 5 (5) | 0 (0)
Headache (Nervous system disorders) | 8 (9) | 4 (4)
Hypertension (Vascular disorders) | 17 (19) | 2 (2)
Flushing (Vascular disorders) | 1 (1) | 2 (2)
Sleep Apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 5 (6) | 0 (0)
Chills (General disorders) | 1 (1) | 2 (2)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 4 (4) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 5 (6) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Peyronie's disease (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Lower urinary tract symptoms (Renal and urinary disorders) | 0 (0) | 2 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-02-18): https://cdn.clinicaltrials.gov/large-docs/28/NCT03198728/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-28): https://cdn.clinicaltrials.gov/large-docs/28/NCT03198728/SAP_001.pdf